CLINICAL TRIAL: NCT04757883
Title: Immunological Follow-up After COVID 19 Vaccination in Kidney Transplant Recipients
Brief Title: Immunological Follow-up After SARS CoV2 Vaccination in Kidney Transplant Recipients
Acronym: COVATRHUS
Status: Terminated | Type: Observational
Why Stopped: the required number of patients has been reached
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8135
Record Dates: First submitted 2021-02-11; First posted 2021-02-17 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Kidney Transplant Recipients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Study of the synthesis of antibodies directed against SARS — Between 5 mL and 45 mL of additional blood will be collected to study the synthesis of antibodies against CoV-2 SARS and to investigate whether specialised immune cells also show an effective response against the virus.

SUMMARY:
The investigators goal is to assess the vaccine response of kidney transplant patients following vaccination against SARS-CoV-2.

The study population will be derived from cohorts of kidney transplant patients who have been transplanted for more than 3 months and have no contraindications to vaccination. These patients will be vaccinated as part of routine care with a CoV-2 SARS vaccine licensed in France.

In this cohort, the investigators wish to study the post-vaccination humoral response by assaying neutralizing antibodies against SARS CoV-2 and the specific cellular response of SARS Cov-2 by quantiferon and in vitro lymphocyte stimulation assays.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older
* Patient vaccinated against SARS-CoV-2 as part of routine care
* Kidney or pancreatic kidney transplant
* Transplantation for more than 3 months
* Subject affiliated to a social protection health insurance
* Subject able to understand the objectives and risks of the research and to give signed and dated informed consent

Exclusion Criteria:

* History of anaphylactic shock or known allergy to PEG
* Known history of COVID or positive Covid serology in the 3 months prior to vaccination
* Contraindication to an intramuscular injection
* Impossibility to give informed information about the subject (subject in an emergency situation, difficulties in understanding the subject, ...)
* Subject under safeguard of justice
* Subject under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: kidney transplants
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the rate of kidney transplant patients with neutralizing Antibodies directed against the Spike protein of the SARS CoV-2 virus after the 2nd injection of the vaccine. | Month 1 after vaccination
The primary endpoint will be the rate of kidney transplant patients with neutralizing Antibodies directed against the Spike protein of the SARS CoV-2 virus after the 2nd injection of the vaccine. | Month 3 after vaccination
The primary endpoint will be the rate of kidney transplant patients with neutralizing Antibodies directed against the Spike protein of the SARS CoV-2 virus after the 2nd injection of the vaccine. | Month 6 after vaccination
The primary endpoint will be the rate of kidney transplant patients with neutralizing Antibodies directed against the Spike protein of the SARS CoV-2 virus after the 2nd injection of the vaccine. | Month 12 after vaccination
The primary endpoint will be the rate of kidney transplant patients with neutralizing Antibodies directed against the Spike protein of the SARS CoV-2 virus after the 2nd injection of the vaccine. | Month 24 after vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Caillard Sophie, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided